CLINICAL TRIAL: NCT04381117
Title: A Phase 2b, Open-label Long-term Durability Study of CCH Following Treatment of Edematous Fibrosclerotic Panniculopathy (Cellulite)
Brief Title: Long-term Durability Study of Collagenase Clostridium Histolyticum (CCH)
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EN3835-220
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Edematous Fibrosclerotic Panniculopathy
Keywords: EFP; Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Treatment: Subjects who participated in and completed study EN3835-201 and had composite improvement of at least 2-levels on both the Clinician Reported-Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient Reported-Photonumeric Cellulite Severity Scale (PR-PCSS) in EN3835-201 study will be eligible for this study. The study will consist of a single day evaluation approximately 4 years after the first dose of the study drug was received in the EN3835-201 study.
  Interventions: Drug: Previously Treated with EN3835

INTERVENTIONS:
Drug: Previously Treated with EN3835 — No treatment to be administered - Observational only

SUMMARY:
This study will evaluate the long-term safety and duration of efficacy of CCH in the treatment of women with cellulite. This study will be a single day evaluation, approximately 48 months after the first dose of study drug was received in the EN3835-201.

ELIGIBILITY:
Inclusion Criteria:

1. Have participated in and completed studies EN3835-201, EN3835-202 and EN3835-219 and had composite improvement of at least 2 levels on both the CR-PCSS and PR-PCSS in study EN3835-201.
2. Be willing and able to cooperate with the requirements of the study.

Exclusion Criteria:

1. Has had retreatment with CCH in the area initially treated during the EN3835-201 study since the completion of study EN3835-219.
2. Has received collagenase treatments (eg, Santyl® Ointment and/or Xiaflex®/Xiapex®) since the completion of study EN3835-219.
3. Has had liposuction on the body region treated during the EN3835-201 study since the completion of that study.
4. Has had any surgery, invasive procedure (eg, liposuction), injectable treatment (eg, KYBELLA®) or any similar treatment in the area treated during the EN3835-201 study since the completion of that study.
5. Has any other condition(s) that, in the investigator's opinion, might indicate the participant to be unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The Durability Population, defined as all subjects in the Safety Population who have both CR-PCSS and PR-PCSS assessments at Visit 1 (Month 48).
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
CR-PCSS change from baseline (Day 1) and reference time point (Day 71) from the EN3835-201 study | Approximately 4 weeks
  Clinician Reported-Photonumeric Cellulite Severity Scale is a 5-level photonumeric scale with ratings ranging from 0 (None) to 4 (Severe)
PR-PCSS change from baseline (Day 1) and reference time point (Day 71) from the EN3835-201 study | Approximately 4 weeks
  Patient Reported-Photonumeric Cellulite Severity Scale is a 5-level photonumeric scale with ratings ranging from 0 (None) to 4 (Severe)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chajko, Study Director — Endo Pharmaceuticals
Locations (4):
- United States (4):
  - Clinical Trial Site #4, Clearwater, Florida
  - Endo Clinical Trial Site #2, Coral Gables, Florida
  - Endo Clinical Trial Site #3, Washington, Missouri
  - Endo Clinical Trial Site #1, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP